CLINICAL TRIAL: NCT01866449
Title: Prospective Controlled Phase 2 Trial of Cabazitaxel in Patients With Temozolomide Refractory Glioblastoma Multiforme (GBM)- The C-GBM Study -
Brief Title: Prospective Phase 2 Trial of Cabazitaxel in Patients With Temozolomide Refractory Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Lars Bullinger, Prof. Dr. med., University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-GBM (XRP6258)
Record Dates: First submitted 2013-05-22; First posted 2013-05-31 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Glioblastoma Multiforme (GBM) WHO Grade IV
MeSH Terms: conditions — Glioblastoma | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental): Cabazitaxel will be given at a dose of 25mg/m² as 1h infusion every 3 weeks
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel
  Other Names: Jevtane

SUMMARY:
The proposed study is an open-label, single-arm, Phase- II trial to assess the efficacy of cabazitaxel in GBM WHO grade IV patients with a progression during or within 6 months after last temozolomide treatment (Figure 1).

Cabazitaxel will be given at a dose of 25mg/m² as 1h infusion every 3 weeks with standard concomitant medication (as outlined below):

* On Day 1 of each cycle, patients will receive cabazitaxel at a dose of 25mg/m², administered by i.v. route in 1 hour.
* Cycle length for cabazitaxel is 3 weeks (21 days).
* New cycles of therapy may not begin until Absolute Neutrophil Count (ANC) ≥1500/mm3, platelet count ≥75 000/mm3, and non-hematological toxicities (except alopecia) have recovered to baseline.
* A maximum of 2 weeks (14 days) delay is allowed between 2 treatment cycles.
* Patients should come off treatment if treatment delay is more than 2 weeks.

At least 30 minutes prior to each administration of cabazitaxel, patients will receive i.v. premedication including:

* An antihistamine (dexchlorpheniramine 5mg, diphenhydramine 25mg, or equivalent). In case of i.v. antihistamine other than promethazine is not being available, local practice should be followed.
* Corticosteroid (dexamethasone 8mg or equivalent)
* H2 antagonist (ranitidine or equivalent).
* Antiemetic prophylaxis is recommended and can be given orally or intravenously if necessary.
* Primary prophylaxis with Granulocyte Colony-Stimulating Factor (G-CSF) should be given on day 4 of each treatment cycle as per ASCO and ESMO guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Both female and male patients meeting the mentioned inclusion and exclusion criteria will be included in this clinical trial. Patients must meet ALL of the following inclusion criteria to be eligible for enrollment into the study:

  * Patients with diagnosis glioblastoma multiforme (GBM) WHO grade IV (histologically confirmed by a pathologist)
  * Progression during or within 6 months after last temozolomide treatment
  * Time since last temozolomide > 21 days
  * Prior external beam radiotherapy (54 to 62 Gy), no option for subsequent radiotherapy
  * No clinical and radiological signs of intracerebral inflammation (in pre-study MRI not older than 4 weeks)
  * Patients > 18 years of age.
  * ECOG performance status of ≤ 2 (stable over 4 weeks prior to study entrance)
  * Female patients of childbearing potential with a negative pregnancy test within 7 days of initiation of study treatment. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
  * Male and female patients of reproductive potential who agree to employ an effective method of birth control throughout the study and for up to 6 months following discontinuation of study drug.
  * Signed informed consent prior to initiation of any study procedure (Must understand, voluntarily sign the informed consent form and be able to adhere to the study visit schedule and other protocol requirements.)

Exclusion Criteria:

* The presence of ANY of the following criteria will exclude a patient from study enrollment:

  * Female patients who are pregnant or breast-feeding
  * History of severe hypersensitivity reaction (≥grade 3) to any component of the investigational drugs or excipients (allergy to or other intolerability of gadolinium, docetaxel, cabazitaxel or polysorbate 80 containing drugs)
  * Unable to undergo Gd-MRI
  * Time since external beam radiotherapy <12 weeks
  * Patients who have been treated with any investigational agent(s) within 28 days of the first day of administration of study drug.
  * Current active second malignancy other than non-melanoma skin cancers and post-treatment of localized prostate cancer. Patients are not considered to have a currently active malignancy if they are in complete remission for > 3 years prior to study
  * Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
  * Known HIV infection, active Hepatitis B or C infection
  * Any serious and/or unstable pre-existing psychiatric or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
  * Any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity (except alopecia) and delayed hematological recovery following last temozolomide cycle
  * Additional anti-cancer treatment for GBM other than study drug and supportive measures (i.e. dexamethasone)
  * Inadequate organ and bone marrow function as evidenced by:

    1. Hemoglobin <9.0 g/dL
    2. Absolute neutrophil count <1.5 x 109/L,
    3. Platelet count <100 x 109/L,
    4. AST/SGOT and/or ALT/SGPT >1.5 x ULN;
    5. Total bilirubin >1.0 x ULN,
    6. Serum creatinine >1.5 x ULN. If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance <60 mL/min should be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Response including SD, PR or CR determined by MRI (modified RANO criteria) | 1 year
  • Response after 12 weeks

SECONDARY OUTCOMES:
Overall and progression-free survival | 3 years
Safety and tolerability | 3 years
  * Rates of deaths within 12 weeks
  * Hematological and non hematological toxicity grade ≥ 2 according to CTCAE V4.0
Pharmacokinetics data concerning drug interactions (i.e. CYP3A induction) | 3 years
  Pharmacokinetics of cabazitaxel in patients with and without concomitant anticonvulsive medication with respect to induction of CYP3A
Quality of life and neurocognitive functioning | 3 years
  Assessment of quality of life, determined by assessment with EORTC QLQ questionnaires (C30 and BN20), and neurocognitive functioning, determined by repeated standardized measurements using MMSE

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Hämatologisch onkologische Praxis, Augsburg
  - Stiftungsklinikum Mittelrhein GmbH, Koblenz
  - Lars Bullinger, MD, Ulm